CLINICAL TRIAL: NCT04754984
Title: A Randomized Trial: Can a Postpartum Pelvic Floor Education Workshop in a High-Risk Population Improve Pelvic Floor Symptoms?
Brief Title: Postpartum Pelvic Floor Workshop
Acronym: PPFW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hamilton Health Sciences Corporation (Other)
Responsible Party: Principal Investigator, Ola Malabarey, Gynecologist, Urogynecology speciality, Hamilton Health Sciences Corporation
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-10672
Record Dates: First submitted 2021-02-09; First posted 2021-02-15 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Pelvic Floor Disorders; Pelvic Floor; Incompetency; Pelvic Floor Muscle Weakness; Perineum; Injury
Keywords: postpartum perineal education
MeSH Terms: conditions — Pelvic Floor Disorders; Wounds and Injuries

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to the intervention or control group. The intervention group will receive the perineal education workshop. The control group will receive standard care. Both groups will receive surveys at baseline, 3, 6 and 12 months postpartum to assess pelvic floor distress.
Masking Description: No masking is possible due to the nature of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): One-time in-person workshop with pelvic floor physiotherapist
  Interventions: Behavioral: Pelvic floor workshop
- Control (No Intervention): Standard care

INTERVENTIONS:
Behavioral: Pelvic floor workshop — Physiotherapist-led workshop on managing pelvic floor symptoms
  Arms: Intervention

SUMMARY:
After having a baby, there are some expected changes in pelvic floor function. However, tearing of the pelvic floor, having a large baby and needing a vacuum or forceps to deliver the baby put women at risk for having pelvic floor disorders. Our study aims to see if, in women who had a high risk for pelvic floor disorders, a pelvic floor education workshop four weeks after delivery can improve pelvic floor disorders compared to those that did not have a workshop.

DETAILED DESCRIPTION:
There is compelling evidence for the need for perineal education and care, especially in women who have recognized risk factors. For example, 30-50% of women who have a clinically recognized risk factor report anal incontinence, fecal urgency, dyspareunia and perineal pain. Despite this, a study found that less than 50% of women with anal incontinence voice those symptoms unless directly asked about them.

Some authors discuss how women may not share these symptoms with their care providers out of the belief that it is a "normal" effect of childbirth. A review of the literature shows that antenatal educational workshops can be an effective means to provide pregnant women with information regarding pelvic floor health, including how modes of delivery impact pelvic floor function. Similarly, antenatal pelvic floor workshops have been found to improve patients' knowledge on pelvic floor health, their practice of pelvic floor muscle exercises and their confidence with these exercises.

To our knowledge, there is no literature exploring the role of a postpartum pelvic floor workshop, on managing perineal and pelvic floor symptoms in women who are identified as being at higher risk of developing pelvic floor dysfunction. Our goal is to develop and assess such a workshop.

ELIGIBILITY:
Inclusion Criteria:

* Postpartum (ie no more than 4 weeks postpartum at time of group allocation)
* Vaginal delivery
* Sustained one or more of the following insults to perineum/pelvic floor

  * Third or fourth degree laceration
  * Vacuum or forceps assisted vaginal delivery
  * Delivery of macrosomic infant ≥4000g)

Exclusion Criteria:

* Prior pelvic floor physiotherapy treatment
* Prior surgical management for pelvic organ prolapse or incontinence
* Unable to understand English
* Caesarean delivery
* Concerns for patient sensitivity - eg if team is aware of neonatal demise, neonate unwell in NICU etc

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2023-03-20 (Actual); Study Completion 2023-03-20 (Actual)

PRIMARY OUTCOMES:
Pelvic floor distress inventory | Differences between groups in the change in score from beginning of study to 3 months post-partum
  Survey on symptoms of pelvic floor distress
Pelvic floor distress inventory | Differences between groups in the change in score from beginning of study to 6 months post-partum
  Survey on symptoms of pelvic floor distress
Pelvic floor distress inventory | Differences between groups in the change in score from beginning of study to 12 months post-partum
  Validated survey on symptoms of pelvic floor distress

SECONDARY OUTCOMES:
Adherence to pelvic floor exercises | From beginning of study to 12 months post-partum
  Investigator generated questions; Difference between groups in proportion who reported adherence to pelvic floor exercises
Seeking medical care for pelvic floor symptoms | from beginning of study to 12 months post-partum.
  Investigator generated questions: Difference between groups in proportion who reported seeking medical care for their symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Ola Malabarey, Principal Investigator — Hamilton Health Sciences, McMaster University
Locations (2):
- Canada (2):
  - Hamilton Health Sciences, Hamilton, Ontario
  - St. Joseph's Healthcare Hamilton, Hamilton, Ontario

IPD SHARING:
Plan to Share IPD: No
There is no place to share IPD with other researchers